CLINICAL TRIAL: NCT07375537
Title: FLIGHT - Autism: An Open-Label, Prospective Study Evaluating the Feasibility and Effectiveness of an Education and Health Coaching Program Focused on Modifiable Lifestyle Factors for Parents of Children With Newly Diagnosed Autism
Brief Title: FLIGHT - Autism: Education and Health Coaching Program Focused on Modifiable Lifestyle Factors for Parents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Documenting Hope Project (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DH-002
Record Dates: First submitted 2026-01-14; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Autism
Keywords: Autism; Environmental modifications; Modifiable lifestyle factors; Parent coaching; Parent education
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parent education and coaching program for newly diagnosed autism (Experimental): Education and coaching program for parents of children with newly diagnosed autism focused on modifiable lifestyle factors and environmental modifications
  Interventions: Behavioral: Parent education and coaching program for newly diagnosed autism

INTERVENTIONS:
Behavioral: Parent education and coaching program for newly diagnosed autism — Education and coaching program for parents of children with newly diagnosed autism that is focused on modifiable lifestyle factors and environmental modifications.

SUMMARY:
The primary purpose of this study is to evaluate the feasibility and effectiveness of an education and coaching program for parents of children with newly diagnosed autism that is focused on modifiable lifestyle factors and environmental modifications. A single-arm, open-label, prospective study will be conducted evaluating the feasibility and effectiveness of the 12-month education and health coaching intervention for parents as an adjuvant to comprehensive clinical care for 12 newly diagnosed children with autism.

ELIGIBILITY:
Inclusion Criteria:

1. Child from 3-7 years of age
2. Child has autism diagnosis (score on the Autism Diagnostic Observation Schedule, 2nd Edition [ADOS-2] ≥ 7) within the last 12 months
3. Child has an Autism Treatment Evaluation Checklist (ATEC) score at screening of between 50 and 79 (considered Level II autism requiring substantial support)
4. Child and parents live in the United States
5. Parent has ability to speak and read English
6. Parents are willing to fulfill study expectations
7. Child has not yet engaged in comprehensive diet, lifestyle, and environmental interventions for autism

Exclusion Criteria:

1. Parents who are unwilling or unable to make lifestyle changes, such as significant dietary changes
2. Parents who are unwilling or unable to participate in study activities, such as group and individual coaching
3. Parents who hold beliefs that are incompatible with an education and lifestyle intervention
4. Child who requires significant specialty medical care, including routine or frequent in-patient medical treatment, are currently taking mood stabilizing drugs, and/or who have cancer or a pre-cancerous condition
5. Child who has been diagnosed with complex conditions in addition to autism, such as an inborn error of metabolism identified through genetic testing, or a known chromosomal disorder
6. Parents who are unable or unwilling to provide consent

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Autism Treatment Evaluation Checklist (ATEC) | Assessed at baseline, six months, 12 months
  The assessment consists of four subtests: Speech/Language Communication (14 items), Sociability (20 items), Sensory/Cognitive Awareness (18 items), and Health/Physical/Behavior (25 items). Each item is rated on a scale from 0 (no problem) to 3 (severe problem), with total scores ranging from 0 to 180. Lower scores indicate less autism symptom severity.

SECONDARY OUTCOMES:
Behavior Assessment System for Children, Third Edition (BASC-3) | Assessed at baseline, 6 months, and 12 months
  Score range: 0 to 100. Interpretation: Lower scores indicate fewer problematic behaviors.
Short Sensory Profile 2 | Assessed at baseline, 6 months, and 12 months
  Raw scores are converted to percentiles. Lower scores indicate fewer sensory behaviors.
Children's Sleep Habits Questionnaire (CSHQ) | Assessed at baseline, 6 months, and 12 months
  Score range 45-135. Lower scores indicate less sleep disturbance.
Goodenough Assessment of Child Drawing | Assessed at baseline, 6 months, and 12 months
  Scores range from 40 to 160. Higher scores indicate greater developmental level.
Autism Diagnostic Observation Schedule, Second Edition (ADOS-2) | Assessed at baseline and 12 months
  Calibrated severity scores range from 1-10. Lower scores indicate lower autism symptom severity.
Automated Self-Administered 24-hour Dietary Assessment Tool (ASA-24) | Assessed at baseline, 6 months, and 12 months.
  No single summed score, as food intake is assessed without maximums or minimums. Lower intake of ultraprocessed foods is the desired outcome.

OTHER OUTCOMES:
Parenting Stress Index-Short Form (PSI-SF) | Assessed at baseline, 6 months, and 12 months.
  Total scores range from 36-180. Lower scores indicate less parental stress.
Quick Environmental Exposure and Sensitivity Inventory (QEESI) | Assessed at baseline, 6 months, and 12 months.
  Scores range from 0-100 for each scale. Lower scores indicate less severe symptoms.
Environmental toxin and functional laboratory panel | Assessed at baseline, 6 months, and 12 months
  Exploratory analysis of environmental toxin and functional laboratory panel. Higher levels indicate worse environmental toxin and functional status. A composite toxin burden ("low", "medium", "high") will be assessed across the panel.

IPD SHARING:
Plan to Share IPD: No
This study of outcomes among children with autism represents a vulnerable population.